CLINICAL TRIAL: NCT06893250
Title: Orthobiologic Treatment for Knee Osteoarthritis (Ortobiologisk Behandling av Kneleddsartrose)
Brief Title: Orthobiologic Treatment for Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 376638
Record Dates: First submitted 2024-10-02; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis Knee
Keywords: osteoarthritis; knee; platelet rich plasma; adipose tissue
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Platelet rich plasma (PRP) (Active Comparator): Plasma taken from the patient is centrifuged and isolated before it is injected into the patients knee.
  Interventions: Biological: PRP injection
- Adipose tissue stem cells (Active Comparator): Adipose tissue is taken from the patients abdominal subcutaneous fat tissue and is injected into the knee.
  Interventions: Biological: ADSTEM Inj. (Adult human mesenchymal stem cells)
- Platelet rich plasma + adipose tissue stem cells (Active Comparator): A combination of platelet rich plasma and adipose tissue stem cells are taken from the patient and injected into the patients knee.
  Interventions: Biological: Injection
- Placebo (saline) (Placebo Comparator): Saline (NaCl) is injected into the patients knee.
  Interventions: Biological: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Biological: PRP injection — Platelet rich plasma, blood from the patient that is centrifuged.
  Other Names: Platelet rich plasma; PRP
  Arms: Platelet rich plasma (PRP)
Biological: ADSTEM Inj. (Adult human mesenchymal stem cells) — Adipose tissue stem cells, from abdominal fat.
  Other Names: Mesenchymal stem cells; Adipose tissue stem cells
  Arms: Adipose tissue stem cells
Biological: Injection — PRP + adipose tissue stem cells
  Other Names: PRP; Adipose tissue stem cells
  Arms: Platelet rich plasma + adipose tissue stem cells
Biological: Saline (NaCl 0,9 %) (placebo) — Sterile saline injection.
  Other Names: placebo; NaCl; saline
  Arms: Placebo (saline)

SUMMARY:
The goal of this randomized clinical trial is to compare treatment for osteoarthritis in the knee using platelet rich plasma (PRP) or adipose stem cells (ADS). The main questions it aims to answer are:

* Will the patients clinically benefit from the treatment, and if so, which treatment is better?
* Will there be radiological findings to support this? Participants will be randomized into one of four groups: PRP, ADS, PRP + ADS or placebo treatment (saline) and will be examined and get an X-ray and MRI of the knee taken at inclusion and after 1 and 2 years.

DETAILED DESCRIPTION:
Patients will be randomized into one of four treatment groups and then be followed up at 6 weeks, 12 weeks, 6 months, 1 year and 2 years after intervention. They will fill out scores and be clinically evaluated, as well as radiologically examined at inclusion and at the final check up (x-ray and MRI).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis in the knee grade I-III using the Kellgren-Lawrance Grading Scale
* Age 40-70 years
* Minimum VAS 3
* No use of NSAIDs or steroids the last 14 days
* No injections of hyaluronic acid the last three months
* Varus/valgus deformity <5 degrees as evaluated on x-ray imaging

Exclusion Criteria:

* Pregnant or breastfeeding women
* Cancer
* Other etiologies of knee pain (refered pain, pain from the back, dislocated meniscus on MRI, osteoarthritis grade IV using the Kellgren-Lawrance Grading Scale)
* Previous knee surgery on the affected knee
* Secondary osteoarthritis in the knee
* Previous infection in the knee
* Other diseases (rheumatoid arthritis, diabetes, systemic diseases or corticosteroid-demaning disease)
* Patients with a high risk of deep vein thrombosis
* Patients who cannot cooperate/are low compliance (psychiatric disease) or has contraindications for MRI

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
KOOS (The Knee injury and Osteoarthritis Outcome Score) | Evaluated during 2 years of follow up (6 weeks, 12 weeks, 6 months, 1 year, 2 years)
  KOOS score filled out by the patient, from 0-100 where a higher score indicates worse outcomes.
WOMAC score (Western Ontario og McMaster Universities Osteoarthritis Index) | Evaluated during 2 years of follow up (6 weeks, 12 weeks, 6 months, 1 year, 2 years)
  Clinical outcome scores (WOMAC) filled out by the patient. Scale from 0-96 in total (0-4 on each question, added together). A higher score indicates a worse score.
VAS (Visual analogue scale) | Evaluated during 2 years of follow up (6 weeks, 12 weeks, 6 months, 1 year, 2 years)
  Pain score (VAS) from 0-10 where a higher score indicates worse outcomes.

SECONDARY OUTCOMES:
Radiological findings after treatment | At inclusion and 2 years after intervention.
  Cartilage status on MRI (magnetic resonance imaging) 2 years after intervention as compared with at time of inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital in Northern Norway, Tromsø, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
Only main scientists in the project will have access to IPD.